CLINICAL TRIAL: NCT01232101
Title: Covered and Uncovered Self Expandable Metallic Stents Are Equally Efficacious in Bile Duct Strictures. Results of a Randomized Study.
Brief Title: Covered or Uncovered Bile Duct Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUMS-01
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Bile Duct Neoplasms
Keywords: covered, uncovered, palliative treatment, stent
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- covered self expandable metallic stents (Active Comparator): Patients with bile malignant bile duct strictures are randomized to covered or uncovered stent
  Interventions: Device: covered or uncovered stents
- Uncovered self expandable metallic stent (Active Comparator)
  Interventions: Device: covered or uncovered stents

INTERVENTIONS:
Device: covered or uncovered stents — Patients are randomized to covered or uncovered stent. Stent patency is monitored and compared as well as complications, efficacy and technical success.
  Other Names: ERCP; Bile duct neoplasms

SUMMARY:
The study is investigator initiated. Tumors that gives the narrowing of the bile ducts prevents bile from flowing from the liver to the intestine resulting in jaundice and the risk of bacterial growth in bile with severe infections as a result. Unresectable bile duct strictures have routinely been treated them with plastic stents. The plastic stents have been replaced by self expandable metallic stents.

These stents remain open longer for reasons that they have a larger diameter so that the bile flows through more easily. One problem with these stents, however, is that the tumor growing through the wire mesh which forms the wall of the stent. This has led to the development of so-called covered stents. Whether covered stents have longer patency is unclear as well as whether they are as safe. There is reason to believe that covered stents remain open longer, but there may be an increased risk of migration and other complications.

The purpose is to prospectively and randomized compare the two stent types. The study endpoint is the clogging of the stent or the patient's death. We also monitor complications, regress time of the jaundice and success rate of stent placement

DETAILED DESCRIPTION:
0

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable, distal bile duct stricture needing relieved endoscopically
* Expected survival greater than 3 months
* The patient must give written consent to participate in the study

Exclusion Criteria:

* Stricture close to hilus
* Need for interpreter

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary aim of the present study was to compare and stent patency between covered and uncovered bileduct SEMS | Stent occlusion or patient death

SECONDARY OUTCOMES:
Secondary objectives were to study difference in technical success, efficacy of drainage and complication rate between covered and uncovered metal stents | Evaluated within three days

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Arne Ung, PhD, MD, Study Director — Dpt Int Med, Skovde
Locations (1):
- Kjell-Arne Ung, Dpt of Internal Medicine, Karnsjukhuset,, Skövde, Sweden